CLINICAL TRIAL: NCT00047840
Title: A Randomized, Double-blind, Multicenter, Phase II Study to Assess the Safety, Tolerability, and Efficacy of ZD6474 in Combination With Docetaxel (TAXOTERE™) in Subjects With Locally Advanced or Metastatic Non-small Cell Lung Cancer (NSCLC) After Failure of Prior Platinum-based Chemotherapy.
Brief Title: This Study is to Assess the Efficacy and Safety of ZD6474 in Subjects With Non-small Cell Lung Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6474IL/0006; NCT00054093 (obsolete NCT alias)
Record Dates: First submitted 2002-10-18; First posted 2002-10-24 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC, Locally Advanced or Metastatic, Second-line
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — vandetanib; Docetaxel

INTERVENTIONS:
Drug: ZD6474
Drug: Placebo
Drug: Docetaxel

SUMMARY:
The purpose of this study is to assess the efficacy and safety of ZD6474 in patients with NSCLC after Failure of Prior Platinum-based Chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic confirmation of NSCLC (locally advanced or metastatic, IB-IV)
* Failure of first-line platinum-based chemotherapy

Exclusion Criteria:

* Mixed small cell or non-small-cell histology
* Bronchoalveolar carcinoma
* Prior chemotherapy or herbal preparations must be discontinued more than 4 weeks before the start of study therapy (6 weeks for nitrosoureas, mitomycin and suramin)
* Prior treatment with docetaxel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129
Dates: Start 2002-10; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Outcome Progression free survival

SECONDARY OUTCOMES:
Incidence and type of adverse events (Aes), clinically significant laboratory abnormalities, and ECG changes;
Objective response rate and duration of response
QoL and lung cancer subscale (LCS) from the FACT-L questionnaire
WHO performance status
Time to death

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (26):
- United States (16):
  - Research Site, Los Angeles, California
  - Research Site, Jacksonville, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, New Orleans, Louisiana
  - Research Site, Boston, Massachusetts
  - Research Site, Pittsfield, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, Billings, Montana
  - Research Site, Great Neck, New York
  - Research Site, New York, New York
  - Research Site, Durham, North Carolina
  - Research Site, Coos Bay, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Houston, Texas
- Czechia (6):
  - Research Site, Brno
  - Research Site, Chomutov
  - Research Site, Hradec
  - Research Site, Ostrava
  - Research Site, Pilsen
  - Research Site, Prague
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Deszk
  - Research Site, Törökbálint